CLINICAL TRIAL: NCT00487266
Title: Soft Tissue Biomechanical Behavior During Acupuncture in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Helene M. Langevin, Professor, National Center for Complementary and Integrative Health (NCCIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01AT003479-01A1 (NIH); 07-025 (Other: CHRMS)
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Low Back Pain
Keywords: Acupuncture; Torque; Force Decay
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Acupuncture — Acupuncture of low back and legs.

SUMMARY:
The goal of this proposal is to test the overall hypothesis that subjects with chronic or recurrent low back pain have an abnormal soft tissue response to acupuncture needling, and that this altered response is associated with abnormal perimuscular connective tissue structure and biomechanics. We will also test whether or not altered needling responses in low back pain are generalized, or localized to specific locations as predicted by traditional acupuncture theory. This proposal is part of a series of projects investigating the role of connective tissue in the mechanism of acupuncture and, in addition, constitutes a first step in examining the role of connective tissue in low back pain. Acupuncturists describe qualitatively different needling responses at locations believed to be "involved" in the patient's disease process. Although assessing abnormalities in the needling response is a fundamental aspect of acupuncture therapy, what constitutes a normal vs. abnormal needling response has never been studied quantitatively. Thus the nature of tissue changes underlying these phenomena remains unknown. We have recently developed a new in vivo technique based on ultrasound elastography that allows visualization and quantification of tissue displacement and strain patterns developed in tissues during needle manipulation in humans [1] (Appendix A). In this proposal, we will use ultrasound elastography, ultrasound image analysis and biomechanical modeling to perform 1) quantitative measurement of soft tissue behavior during needling and 2) detailed analysis of perimuscular connective tissue structure and biomechanics in human subjects with and without low back pain.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for LBP subjects will be the following:

1. History of recurrent or chronic LBP as defined by Von Korff {Von Korff, 1992 #6777} {Von Korff, 1994 #6816} for a minimum of 12 months
2. Able to stand and walk without assistance
3. Able to understand and read English
4. Able to understand and sign a consent form. Subjects' LBP will be further defined as being recurrent or chronic LPB based on the number of days with symptoms over a period of one year.

   * Recurrent LBP will be defined as back pain present on less than ½ the days in a 12-month period, occurring in multiple episodes over a year.
   * Chronic LBP will be defined as back pain present on at least ½ the days in a 12-month period in a single or multiple episodes.

Inclusion criteria for No-LBP subjects:

Criteria for selecting No-LBP subjects will be:

1. No history of low back pain or any other chronic pain that has limited activities of daily living or work
2. A numerical current pain index of less than 0.5. No-LBP subjects will be matched for age, sex and subcutaneous tissue thickness with LBP subjects.

Exclusion Criteria:

For all subjects, exclusion criteria determined by history and physical exam will be the following:

1. Previous severe back or low extremity injury or surgery
2. Major structural spinal deformity (scoliosis, kyphosis, stenosis)
3. Ankylosing spondylitis or rheumatoid arthritis
4. Spondyloarthropathy or disc herniation
5. Spinal fracture, tumor or infection
6. Neurological deficit (weakness and/or sensory loss, decreased deep tendon reflexes suggesting nerve root compression, but not subjective symptoms of nerve root irritation (sciatica)
7. Neurological or major psychiatric disorder
8. Bleeding disorders
9. Corticosteroid or anticoagulant medication
10. Pregnancy
11. worker's compensation or disability case
12. In litigation for the LBP problem
13. Acute systemic infection
14. BMI greater than 23% or less than 32%. Preliminary testing has shown that individuals with a BMI of less than 23% have an insufficient depth of the subcutaneous and fat zone (Zone P) for data processing. Individuals with a BMI greater than 32% have a subcutaneous and fat zone (Zone P) thickness which is greater than the acupuncture needle length, which will not allow penetration of the muscle layer (Zone M).
15. Subjects will need to not take non-steroidal anti-inflammatory (NSAIDs) medication for 3 days prior to testing in order to avoid the potentially confounding acute effects of NSAIDs on connective tissue.
16. In addition, LBP subjects will be excluded if they are in an acute flare-up of LBP. Flare-up will be defined as short period (less than one week) when pain is markedly more severe than usual for that individual (at least 5 points above baseline on pain index).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures will be peak torque during needle rotation (Torque); force decay time constant during needle oscillation (ForceDecay) and tissue displacement (Displacement) in Subcutaneous, Perimuscular and Muscle zones during needle oscillation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Helene M. Langevin, M.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States